CLINICAL TRIAL: NCT04172597
Title: A Phase 2 Study of Poziotinib in Patients With EGFR or HER2 Activating Mutations in Advanced Malignancies
Brief Title: A Study of Poziotinib in Patients With Epidermal Growth Factor Receptor (EGFR) or Human Epidermal Growth Factor Receptor 2 (HER2) Activating Mutations in Advanced Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic business decision (unrelated to safety)
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-POZ-203
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Colorectal Cancer; Solid Tumor; Glioblastome Multiforme
Keywords: EGFR activating mutations; HER2 activating mutations; HER2-positive breast cancer; HER2-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms | interventions — Loperamide

STUDY DESIGN:
Intervention Model Description: Each treatment cycle is 28 calendar days in duration. This is a basket study with five distinct cohorts. Eligible patients will be enrolled into the five cohorts concurrently based on tumor type and mutational status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Patients with HER2-positive or HER2-negative BC with a HER2 activating mutation will receive poziotinib 8 milligrams (mg), orally, twice daily (BID) starting on Day 1 of each 28 day cycle for up to 24 months unless there is disease progression, death, intolerable AEs, or another protocol-specified reason for participant withdrawal. Loperamide may be prescribed for the treatment of diarrhea as needed.
  Interventions: Drug: Poziotinib Hydrochloride; Drug: Loperamide
- Cohort 2 (Experimental): Patients with CRC with a HER2 activating mutation will receive poziotinib 8 mg, orally, BID starting on Day 1 of each 28 day cycle for up to 24 months unless there is disease progression, death, intolerable AEs, or another protocol-specified reason for participant withdrawal. Loperamide may be prescribed for the treatment of diarrhea as needed.
  Interventions: Drug: Poziotinib Hydrochloride; Drug: Loperamide
- Cohort 3 (Experimental): Patients with CRC with a HER2 activating mutation will receive poziotinib 8 mg, orally, BID starting on Day 1 of each 28 day cycle for up to 24 months unless there is disease progression, death, intolerable AEs, or another protocol-specified reason for participant withdrawal. Loperamide may be prescribed for the treatment of diarrhea as needed.
  Interventions: Drug: Poziotinib Hydrochloride; Drug: Loperamide
- Cohort 4 (Experimental): Patients with CRC with a HER2 activating mutation will receive poziotinib 8 mg, orally, BID starting on Day 1 of each 28 day cycle for up to 24 months unless there is disease progression, death, intolerable AEs, or another protocol-specified reason for participant withdrawal. Loperamide may be prescribed for the treatment of diarrhea as needed.
  Interventions: Drug: Poziotinib Hydrochloride; Drug: Loperamide
- Cohort 5 (Experimental): Patients with CRC with a HER2 activating mutation will receive poziotinib 8 mg, orally, BID starting on Day 1 of each 28 day cycle for up to 24 months unless there is disease progression, death, intolerable AEs, or another protocol-specified reason for participant withdrawal. Loperamide may be prescribed for the treatment of diarrhea as needed.
  Interventions: Drug: Poziotinib Hydrochloride; Drug: Loperamide

INTERVENTIONS:
Drug: Poziotinib Hydrochloride — The poziotinib drug substance is a hydrochloride salt of poziotinib and is formulated as a tablet for oral administration.
Drug: Loperamide — Loperamide as prescribed by the physician.

SUMMARY:
This is a Phase 2, open-label, multicenter study whose principal objectives are to evaluate the efficacy and safety/tolerability of poziotinib in five cohorts of 30 previously-treated patients each.

DETAILED DESCRIPTION:
The Screening period (Day -30 to Day 1) begins 30 days prior to poziotinib treatment on Day 1 of Cycle 1. Patients must meet all Inclusion/Exclusion Criteria and provide informed written consent prior to study procedures.

The duration of each treatment cycle is 28 days. There will be five patient cohorts. Eligible patients will be enrolled into cohorts concurrently based on EGFR or HER2 exon 20 mutation status.

* Cohort 1: HER2-positive or HER2-negative breast cancer (BC) with a HER2 activating mutation.
* Cohort 2: Colorectal cancer (CRC) with a HER2 activating mutation.
* Cohort 3: Any solid cancer, except non-small cell lung cancer (NSCLC), BC, or CRC with a HER2 activating mutation.
* Cohort 4: Glioblastome multiforma (GBM) with an EGFR activating mutation.
* Cohort 5: Any solid cancer, except NSCLC or GBM with an EGFR activating mutation.

All patients will be treated daily for up to 24 months unless there is disease progression, death, intolerable adverse events (AEs), or another protocol-specified reason for patient withdrawal. After treatment discontinuation, patients will be contacted every 3 months for up to 2 years after the first dose of poziotinib to assess survival.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients must be at least 18 years old.
2. Patients must have histologic or cytologic evidence of a malignant solid cancer that is either advanced or metastatic there must be no available therapy known to confer a reasonable likelihood of clinical benefit.
3. Patients with BC must have a HER2 activating mutation determined by next-generation sequencing (NGS) performed on either tumor or plasma samples and:

   * Immunohistochemistry (IHC) HER2-positive BC that has progressed on trastuzumab, pertuzumab, and trastuzumab emtansine (T-DM1) in the metastatic setting, unless there is recurrent disease within 12 months of adjuvant or neoadjuvant treatment.
   * IHC HER2-negative, estrogen receptor/progesterone receptor (ER/PR)-positive BC that has progressed on or after appropriate first-line endocrine therapy in the metastatic setting.
   * IHC HER2-negative, ER/PR-negative BC that has progressed after first-line treatment (any standard chemotherapy-based regimen) in the metastatic setting.
4. Patients with microsatellite instability-high (MSI-H) CRC must have had appropriate checkpoint inhibitor-based therapy.
5. Patient's tumor must be positive for an EGFR or HER2 mutation based on DNA testing of either tumor tissue or plasma samples. Patients with documented EGFR or HER2 mutations may be identified by local testing from participating sites using next generation sequencing tests. Patient has a solid tumor with at least one of the listed activating mutations:

   * Cohorts 1-3: HER2 Activating Mutations (at least one of the following) Furin-Like/Extracellular. S310F/Y Transmembrane. I655V, V659E, R678Q, V697L Kinase Domain. Exon 20 insertion, T733I, L755X, I767M, D769X, V773M, V777X, L786V, V842I, T862I, L869R.
   * Cohorts 4-5: EGFR Activating Mutations (at least one of the following) Extracellular & Transmembrane: EGFRvIII, R108K, R222C, A289T, P596L, G598V Kinase Domain: Exon 20 insertion, E709X, E709_T710del insD, L718X, G719X, I740_K745dupIPVAIK, I740_K745dup, V742I, L747X, E746_A750del, A750P, S768I, S768I/V769L, S768I/V774M, L833V, V769M, V774M, R831C, R831H, L858R, L861Q, A864V.
6. Patients must have measurable disease.
7. Patients with central nervous system (CNS) metastases must have stable CNS disease and no evidence of growth on imaging for at least 4 weeks following radiation or other locoregional ablative therapy. CNS symptoms must be stable with no requirement for anti-seizure medications and/or > 2 mg/day dexamethasone equivalent, except for patients with GBM (Cohort 4), in whom anti-seizure medications and/or up to 4 mg/day dexamethasone equivalent is allowed.
8. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ -1.
9. Patients must have adequate hematopoietic, renal, and liver functions.

Exclusion Criteria:

1. Patient has an EGFR T790 mutation.
2. Patient has breast or gastric cancer without eligible HER2 mutations (see Inclusion Criteria).
3. Patients with GBM enrolled in Cohort 4 has been treated with an inhibitor of vascular endothelial growth factor (VEGF) inhibitor therapy (e.g., bevacizumab).
4. Patient requires treatment with a medication that is a strong inhibitor or inducer of CYP3A4 or CYP2D6 or has been treated with such medications within 15 days of poziotinib treatment.
5. Patient has ≥ Grade 2 skin disorders (rash), mucositis, or stomatitis within 15 days of poziotinib treatment.
6. Patient has a gastrointenstinal disorder or malabsorption that precludes oral drug treatment.
7. Patient has active liver or biliary tract disease (except for Gilbert's syndrome, asymptomatic biliary stones, liver metastasis, or stable chronic liver diseases).
8. Patient has a history of drug-induced pancreatitis.
9. Patient has a history of interstitial lung disease or pneumonitis.
10. Patient has a history of congestive heart failure Class III/IV according to the New York Heart Association Functional Classification or a serious cardiac arrhythmia requiring treatment.
11. Patient has a high risk of cardiac disease as determined by the Investigator. If patient is deemed to have a high cardiac risk, enrollment may be considered if an echocardiogram (ECHO) or multi-gated acquisition (MUGA) during Screening demonstrates a cardiac ejection fraction >= 50%.
12. Patient has a QTc interval > 470 ms.
13. Patient has a history of another malignancy within the 1 year prior to poziotinib treatment. Patients with the following concomitant neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ (including transitional cell carcinoma, cervical intraepithelial neoplasia, and melanoma in situ), organ-confined prostate cancer with no evidence of progressive disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaba Kokhreidze, MD, Study Director — Spectrum Pharmaceuticals, Inc
Locations (1):
- Pacific Shores Medical Group, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participant was enrolled at 1 site in the United States.
Groups:
- Cohort 1: Participants with human epidermal growth factor receptor 2 (HER2) positive or HER2-negative breast cancer (BC) with a HER2 activating mutation were to receive poziotinib 8 milligrams (mg), orally, twice daily (BID) starting on Day 1 of each 28-day cycle for up to 24 months unless there is disease progression, death, intolerable adverse events (AEs), or another protocol-specified reason for participant withdrawal. Participants were also to receive loperamide 4 mg two to three times a day according to treating physician's instructions.
- Cohort 2: Participants with colorectal cancer (CRC) with a HER2 activating mutation were to receive poziotinib 8 mg, orally, BID starting on Day 1 of each 28-day cycle for up to 24 months unless there is disease progression, death, intolerable AEs, or another protocol-specified reason for participant withdrawal. Participants were also to receive loperamide 4 mg two to three times a day or according to the treating physician's instructions.
- Cohort 3: Participants with solid tumors (except non-small cell lung cancer (NSCLC), BC, or CRC) with a HER2 activating mutation were to receive poziotinib 8 mg, orally, BID starting on Day 1 of each 28-day cycle for up to 24 months unless there is disease progression, death, intolerable AEs, or another protocol-specified reason for participant withdrawal. Participants were also to receive loperamide 4 mg two to three times a day or according to the treating physician's instructions.
- Cohort 4: Participants with glioblastoma (GBM) with epidermal growth factor receptor (EGFR) activating mutation were to receive poziotinib 8 mg, orally, BID starting on Day 1 of each 28-day cycle for up to 24 months unless there is disease progression, death, intolerable AEs, or another protocol-specified reason for participant withdrawal. Participants were also to receive loperamide 4 mg two to three times a day or according to the treating physician's instructions.
- Cohort 5: Participants with solid tumors (except NSCLC or GBM) with EGFR activating mutations were to receive poziotinib 8 mg, orally, BID starting on Day 1 of each 28-day cycle for up to 24 months unless there is disease progression, death, intolerable AEs, or another protocol-specified reason for participant withdrawal. Participants were also to receive loperamide 4 mg two to three times a day or according to the treating physician's instructions.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 0 | 0 | 0 | 0 | 1
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The study was terminated by the Sponsor. Based on the low enrollment number (n=1), no data is reported here to protect and maintain participant privacy/confidentiality.
Groups:
- Cohort 1: Participants with HER2-positive or HER2-negative BC with a HER2 activating mutation were to receive poziotinib 8 mg, orally, BID starting on Day 1 of each 28-day cycle for up to 24 months unless there is disease progression, death, intolerable AEs, or another protocol-specified reason for participant withdrawal. Participants were also to receive loperamide 4 mg two to three times a day according to the treating physician's instructions.
- Cohort 2: Participants with CRC with a HER2 activating mutation were to receive poziotinib 8 mg, orally, BID starting on Day 1 of each 28-day cycle for up to 24 months unless there is disease progression, death, intolerable AEs, or another protocol-specified reason for participant withdrawal. Participants were also to receive loperamide 4 mg two to three times a day or according to the treating physician's instructions.
- Cohort 3: Participants with solid tumors (except NSCLC, BC, or CRC) with a HER2 activating mutation were to receive poziotinib 8 mg, orally, BID starting on Day 1 of each 28-day cycle for up to 24 months unless there is disease progression, death, intolerable AEs, or another protocol-specified reason for participant withdrawal. Participants were also to receive loperamide 4 mg two to three times a day or according to the treating physician's instructions.
- Cohort 4: Participants with GBM with EGFR activating mutation were to receive poziotinib 8 mg, orally, BID starting on Day 1 of each 28-day cycle for up to 24 months unless there is disease progression, death, intolerable AEs, or another protocol-specified reason for participant withdrawal. Participants were also to receive loperamide 4 mg two to three times a day or according to the treating physician's instructions.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The study was terminated by the Sponsor. Based on the low enrollment number (n=1), no data is reported here to protect and maintain participant privacy/confidentiality.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The study was terminated by the Sponsor. Based on the low enrollment number (n=1), no data is reported here to protect and maintain participant privacy/confidentiality.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The study was terminated by the Sponsor. Based on the low enrollment number (n=1), no data is reported here to protect and maintain participant privacy/confidentiality.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The study was terminated by the Sponsor. Based on the low enrollment number (n=1), no data is reported here to protect and maintain participant privacy/confidentiality.
Region of Enrollment [Number; unit: participants] — Population: The study was terminated by the Sponsor. Based on the low enrollment number (n=1), no data is reported here to protect and maintain participant privacy/confidentiality.

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with confirmed complete response (CR) and partial response (PR) as assessed by the investigator using local radiology evaluation according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1). CR is defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes must have a reduction in the short axis to <10 millimeters (mm). PR is defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR.
Time Frame: Up to 168 days
Population: The Evaluable Population included all enrolled participants who completed at least 6 weeks of poziotinib treatment, had baseline and at least 1 post-baseline tumor response evaluation using RECIST, v1.1, or progressed prior to any post-baseline image evaluation. As the study was terminated early by the sponsor, there were no participants enrolled in cohorts 1-4.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 1: Participants with HER2 positive or HER2-negative BC with a HER2 activating mutation were to receive poziotinib 8 mg, orally, BID starting on Day 1 of each 28-day cycle for up to 24 months unless there is disease progression, death, intolerable AEs, or another protocol-specified reason for participant withdrawal. Participants were also to receive loperamide 4 mg two to three times a day according to treating physician's instructions.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
percentage of participants |  |  |  |  | 0

2. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response was defined as the time from the date that measurement criteria are first met for CR or PR until the first subsequent date that progressive disease or death is documented. CR is defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes must have a reduction in the short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. Disease progression (PD) is defined as ≥20% increase in the sum of diameters of target lesions, unequivocal progression in non-target lesions, and/or appearance of new lesions.
Time Frame: Up to 168 days
Population: The Evaluable Population included all enrolled participants who completed at least 6 weeks of poziotinib treatment, had baseline and at least 1 post-baseline tumor response evaluation using RECIST, v1.1 or progressed prior to any post-baseline image evaluation. As the study was terminated early by the sponsor, there were no participants enrolled in cohorts 1-4.
Groups:
- Cohort 1: Participants with HER2-positive or HER2-negative BC with a HER2 activating mutation were to receive poziotinib 8 mg, orally, BID starting on Day 1 of each 28-day cycle for up to 24 months unless there is disease progression, death, intolerable AEs, or another protocol-specified reason for participant withdrawal. Participants were also to receive loperamide 4 mg two to three times a day according to treating physician's instructions.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as percentage of participants with best response of CR, PR, and stable disease (SD) from the first dose of poziotinib to the end of study. CR is defined as disappearance of all target and non-target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of the longest diameter (LD) since the treatment started.
Time Frame: Up to 168 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
percentage of participants |  |  |  |  | 0

4. Secondary Outcome: Percentage of Participants With AE
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation patient, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Therefore, an AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Time Frame: Up to 30 days after last dose of study drug (Up to 199 days)
Population: The Safety Analysis Population included all enrolled patients who received at least 1 dose of poziotinib. As the study was terminated early by the sponsor, there were no participants enrolled in cohorts 1-4.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
percentage of participants |  |  |  |  | 100

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last dose of study drug (Up to 199 days)
Description: The Safety Analysis Population included all enrolled patients who received at least 1 dose of poziotinib. As the study was terminated early by the sponsor, there were no participants enrolled in cohorts 1-4.
Groups:
- Cohort 1: Participants with HER2 positive or HER2-negative breast cancer (BC) with a HER2 activating mutation were to receive poziotinib 8 mg, orally, BID starting on Day 1 of each 28-day cycle for up to 24 months unless there is disease progression, death, intolerable adverse events AEs, or another protocol-specified reason for participant withdrawal. Participants were also to receive loperamide 4 mg two to three times a day according to treating physician's instructions.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=0) | Cohort 2 (N=0) | Cohort 3 (N=0) | Cohort 4 (N=0) | Cohort 5 (N=1)
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Sinus Tachycardia] (Cardiac disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT04172597/Prot_SAP_000.pdf